CLINICAL TRIAL: NCT05620654
Title: A Phase I Dose-finding Trial of Hyperthermic Intraperitoneal Paclitaxel Combined With Cisplatin in Patients With Advanced-stage Ovarian Cancer
Brief Title: A Phase I Dose-finding Trial of Hyperthermic Intraperitoneal Paclitaxel Combined With Cisplatin
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jing Li, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KY-132
Record Dates: First submitted 2022-11-11; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Ovarian Cancer; Hyperthermic Intraperitoneal Chemotherapy; Paclitaxel
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Intervention Model Description: Bayesian Optimal Interval Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hyperthermic Intraperitoneal Paclitaxel Combined With Cisplatin (Experimental): Patients with ovarian cancer receive hyperthermic intraperitoneal paclitaxel combined with a fixed dose of cisplatin (75mg/m2)
  Interventions: Drug: Hyperthermic Intraperitoneal Paclitaxel Combined With Cisplatin

INTERVENTIONS:
Drug: Hyperthermic Intraperitoneal Paclitaxel Combined With Cisplatin — The starting dose for paclitaxel was 175 mg/m2, with escalation in 25 mg/m2 increments until the MTD was determined or the maximum dose level of 225 mg/m2 was reached. The target dose-limiting toxicity (DLT) rate was 25%, and the total sample size was 30 patients. HIPEC was delivered immediately following the debulking surgery using the closed technique with a target temperature of 43 ℃ for 90 minutes.

SUMMARY:
Primary objective of this trial is to identify the maximum tolerated dose (MTD) of paclitaxel combined with a fixed dose of cisplatin (75 mg/m2) delivered as hyperthermic intraperitoneal chemotherapy (HIPEC) in patients with ovarian cancer.

In this single-center Phase I trial, Bayesian Optimal Interval Design (TITE-BOIN) was used. The starting dose for paclitaxel was 175 mg/m2, with escalation in 25 mg/m2 increments until the MTD was determined or the maximum dose level of 225 mg/m2 was reached. The target dose-limiting toxicity (DLT) rate was 25%, and the total sample size was 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years;
* adequate renal function (blood creatinine: 58-96 µmol/L), bone marrow function (hemoglobin ≥ 110 g/L, white cell count ≥ 4.0 ×109/L, neutrophil count ≥ 2.0 × 109/L, platelet count ≥ 100 × 109/L) and hepatic function [bilirubin 3.4-22.2 µmol/L, alanine aminotransferase (ALT) 7-40 U/L, aspartate aminotransferase (AST) 13-35 U/L, AST/ALT≤ 1.5].

Exclusion Criteria:

* Patients who had been treated with cisplatin OR paclitaxel for any reason within 3 weeks prior to HIPEC.
* A history of HIPEC treatment

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity | within 3 weeks following HIPEC
  Grade 3 AEs according to the National Cancer Institute Common Terminology Criteria for Adverse Event (CTC-AE) Version 4.0 classification are used to define DLT.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: Undecided